CLINICAL TRIAL: NCT06442527
Title: Using Virtual Reality Before Transcranial Magnetic Stimulation for the Treatment of OCD
Acronym: VR-TMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000037937
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: TMS; Transcranial Magnetic Stimulation; Virtual Reality; VR
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): This single arm will include all participants of the study, who will all receive the intervention
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual reality gear and content will be used prior to TMS session as part of the provocation items

SUMMARY:
This study will focus on the use of Virtual Reality (VR) technology in patients receiving treatment using Transcranial Magnetic Stimulation (TMS) for Obsessive-Compulsive Disorder (OCD)

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old
* Patients must have been clinically evaluated by a Yale Interventional Psychiatry Service physician who has deemed them appropriate to receive TMS for the treatment of OCD
* Ability and willingness, in the investigator's judgement, to comply with the study procedure and study requirements.

Exclusion Criteria:

* Hearing or visual impairment to the degree that would interfere with ability to see or hear VR content.
* Difficulty in understanding spoken or written English
* Pregnancy
* History of seizure disorder
* Unable to provide informed consent
* Dementia or other cognitive disorder or intellectual disability that would impair the subject's ability to understand the study procedure (per investigator judgment)
* Any implanted medical device, risk of interference with which by the VR device in the investigator's judgment can put patient at additional undue risk.
* Any other medical or psychiatric comorbidity that the investigator judges would put the participant at additional undue risk due to study participation or would impair subject's ability to participate in the study.
* Was previously enrolled/randomized into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tolerability of VR treatment by qualitative assessment | Within 1 hour after each treatment session
  Tolerability will be assessed by open-ended interview of the patient about their experience and any difficulty tolerating VR

CONTACTS AND LOCATIONS:
Overall Officials: Sina Nikayin, MD, Principal Investigator — Assistant Professor, Departement of Psychiatry, Yale University
Locations (1):
- Yale Psychiatry Hospital Interventional Psychiatry Services (IPS) unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No